CLINICAL TRIAL: NCT06301100
Title: Single-center, Prospective Study on the Identification and Delineation of Brain and Lung Tumors and At-Risk Organs, and Functional Testing of Surrounding Tissues Based on Dual-Energy CT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E20230371
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-04

CONDITIONS: Image Quality and Contouring Accuracy of the Tumor in Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dual energy CT after routine simulation — Dual energy CT after routine simulation

SUMMARY:
This study explored the feasibility of dual-energy CT in head and lung tumors. Dual-energy CT can achieve quantitative CT imaging based on traditional imaging by dual-energy spectral imaging, and enhance the clarity of head and lung tumors. In this study, we will prospectively explore the image accuracy and delineation accuracy of dual energy CT in radiotherapy to verify whether dual energy CT performs better with conventional CT.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in and sign the informed consent in person. 2. Over 18 years old, gender unlimited; 3. After imaging diagnosis of primary lung cancer or space-occupying lung lesions with oligometastases, MDT decided to treat SBRT 4. Clinical stage IA-IV (cT1-4N1-3M0-1); 5. No serious abnormality of blood system, heart, lung, liver, kidney function and immune deficiency; 6. Coagulation function: activated partial thromboplastin time (APTT) < the upper limit of normal 10 seconds, prothrombin time (PT) < the upper limit of normal 3 seconds, plasma fibrinogen 2-4g/L; 7. Hemoglobin ≥100g/L, WBC≥4×109/L, neutrophils ≥1.5×109/L, platelets ≥100×109/L 8. Bilirubin < 1.5 times the upper limit of normal value; Glutamic oxalic aminotransferase (ALT) & Glutamic pyruvic aminotransferase (AST) ≤1.5 times the upper limit of normal value; 9. Serum creatinine ≤1.5 times the upper limit of normal value; 10. The willingness of men or women of childbearing age to use contraception in the trial; 11. Physical condition score ECOG level 0 ~ 2; 12. Expected survival >3 months;13, Can acquire MRI scanning

Exclusion Criteria:

1. Patients could not tolerate or were unwilling to undergo CT examination; 2. The primary lesion has undergone surgery or radiotherapy or chemotherapy or targeted or immunotherapy; 3. Subjects who have received other drug trials within the last 1 month; 4. People with severe allergic history or idiosyncrasies; 5. Patients with a history of severe lung or heart disease; 6. Severe comorbidities, such as uncontrolled hypertension, heart failure, etc.; 7. Pregnant or lactating women; 8. Previous history of malignant tumor; 9. Refusal or inability to sign informed consent to participate in the trial; 10. Currently or planning to participate in other clinical trials; 11,Can not acquire MRI scanning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with primary or metastatic tumors in the lungs and brains, in good general condition and are proposed to undergo SBRT
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-04-28 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
DICE value | 2023.4-2024.12
  The contouring accuracy

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, National Clinical Research Center for Cancer, Key laboratory of Cancer Prevention and Therapy, Tianjin's Clinical Research Center for Cancer, Huan-Hu-Xi, Tianjin, Tianjin Municipality, China